CLINICAL TRIAL: NCT05147493
Title: A Phase 2 Study of Isatuximab in Combination With Bortezomib, Cyclophosphamide and Dexamethasone Followed by Isatuximab and Lenalidomide Maintenance in Newly Diagnosed Patients With Multiple Myeloma and Severe Renal Impairment (EAE116)
Brief Title: A Phase 2 Study of Isatuximab in Combination With Bortezomib, Cyclophosphamide and Dexamethasone Followed by Isatuximab and Lenalidomide Maintenance in Newly Diagnosed Patients With Multiple Myeloma and Severe Renal Impairment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAE116
Record Dates: First submitted 2021-11-05; First posted 2021-12-07 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma; Renal Impairment; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases | interventions — isatuximab; Bortezomib; Cyclophosphamide; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Eligible patients will initially receive an induction phase of six 28-day cycles of Isatuximab in combination with Bortezomib, Cyclophosphamide, and Dexamethasone, followed by a maintenance phase with isatuximab and lenalidomide until disease progression, death, unacceptable adverse events (AEs), lost to follow up, or consent withdrawal, whichever occurs first.
  Isatuximab will be given at a dose of 10 mg/kg once weekly (QW) on Days 1, 8, 15, and 22 in Cycle 1, on Days 1 and 15 during Cycles 2-6 and on Day 1 from Cycle 7 onwards.
  Bortezomib will be given at 1.3 mg/m2 on Days 1, 4, 8, 11 of Cycle 1 and days 1, 8, 15, 22 of Cycles 2-6.
  Cyclophosphamide will be given at 300 mg/m2 on Days 1, 8, 15 of Cycle 1 and days 1, 8, 15, 22 of Cycles 2-6.
  Dexamethasone will be given at 40 mg (20 mg for ≥75 years old) on Days 1-4 and 9-12 of Cycle 1 and Days 1, 8, 15 and 22 of Cycles 2-6.
  Lenalidomide will be given at 10 mg (or according to renal function) daily from Cycle 7 onwards.
  Interventions: Drug: Isatuximab; Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Isatuximab — Route of administration: Intravenous (IV). Dose regimen: Isatuximab will be given at a dose of 10 mg/kg once weekly (QW) on Days 1, 8, 15, and 22 in Cycle 1, on Days 1 and 15 during Cycles 2-6 and on Day 1 from Cycle 7 onwards.
Drug: Bortezomib — Route of administration: Subcutaneous (SC). Dose regimen: Bortezomib will be given at 1.3 mg/m2 on Days 1, 4, 8, 11 of Cycle 1 and days 1, 8, 15, 22 of Cycles 2-6.
Drug: Cyclophosphamide — Route of administration: Intravenous (IV). Dose regimen: Cyclophosphamide will be given at 300 mg/m2on Days 1, 8, 15 of Cycle 1 and days 1, 8, 15, 22 of Cycles 2-6.
Drug: Dexamethasone — Route of administration: per os (PO)/Intravenous (IV). Dose regimen: Dexamethasone will be given at 40 mg (20 mg for ≥75 years old) on Days 1-4 and 9-12 of Cycle 1 and Days 1, 8, 15 and 22 of Cycles 2-6.
Drug: Lenalidomide — Route of administration: per os (PO). Dose regimen: Lenalidomide will be given at 10 mg (or according to renal function) daily from Cycle 7 onwards.

SUMMARY:
This is an Investigator-Initiated, phase 2, prospective, open-label study designed to be conducted in six hospitals in Greece.

Eligible patients will initially receive an induction phase of six 28-day cycles of isatuximab in combination with bortezomib, cyclophosphamide, and dexamethasone (VCd), followed by a maintenance phase with isatuximab and lenalidomide until disease progression, death, unacceptable adverse events, lost to follow up, or consent withdrawal, whichever occurs first. The study will last for approximately 36 months (follow-up period), starting from the date of the first patient in, to the date of the last patient last visit.

The primary objective is to assess the effect of induction treatment with isatuximab in combination with VCd on the renal function of newly diagnosed patients with multiple myeloma and severe renal impairment (RI).

The secondary objectives are to evaluate the effect of isatuximab in combination with VCd, followed by lenalidomide maintenance on: Overall response rate, Progression-Free Survival, Time to Response, Duration of Response, Overall Survival, Minimal Residual Disease negativity rate, Safety

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed an informed consent form (ICF), stating that he or she understands the purpose of the procedures required for the study and is willing to participate in the study. The patient must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as stated in the ICF.
2. Male or female patients aged 18 years or older at the time of the ICF signature.
3. Patients diagnosed with MM based on the International Myeloma Working Group (IMWG) criteria (see Appendix H).
4. Patients with severe RI defined as estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m2 (calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula) or in need for dialysis (see Appendix E).
5. Patients with current evidence of measurable disease defined as:

   * Serum monoclonal protein (M-protein) levels ≥0.5 g/dL, measured using serum protein electrophoresis (SPEP) and/or
   * Urine M-protein levels ≥200 mg/24 hours, measured using urine protein electrophoresis (UPEP), or
   * Serum immunoglobulin free light chain (FLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
6. Adequate bone marrow and hepatic function as defined by ALL the laboratory criteria:

   * Absolute Neutrophil Count (ANC) ≥1.0 x 109/L (Granulocyte colony-stimulating factor (GCSF) administration is not allowed to reach this level)
   * Hemoglobin levels ≥7.5 g/dL (≥4.65 mmol/L)
   * Platelet count ≥75 x 109/L in patients in whom <50% of bone marrow nucleated cells are plasma cells OR platelet count ≥50 x 109/L in patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells (transfusions are not allowed to reach this level)
   * Alanine aminotransferase (ALT) levels ≤2.5 x the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) levels ≤2.5 x ULN
   * Total bilirubin levels ≤1.5 x ULN (except for Gilbert Syndrome: direct bilirubin ≤1.5 x ULN)
   * Serum calcium corrected for albumin ≤14.0 mg/dL (≤3.5 mmol/L), or free ionized calcium ≤ 6.5 mg/dL (≤1.6 mmol/L)
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2 (see Appendix C).
8. For patients experiencing toxicities resulting from previous therapy, the toxicities must be resolved or stabilized to ≤ Grade 1

Exclusion Criteria:

1. Prior or current systemic therapy or stem-cell transplantation for any plasma cell dyscrasia, with the exception of emergency use of a short course (the equivalent of dexamethasone 40 mg/day for a maximum of 4 days) of corticosteroids before treatment.
2. History of malignancy (other than MM) within three years before Cycle 1, Day 1 (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the Investigator, with concurrence with the Sponsor's medical monitor, are considered cured with minimal risk of recurrence within three years).
3. Clinical signs of meningeal involvement of MM.
4. Clinically significant cardiac disease, including:

   1. Myocardial infarction within six months before Cycle 1, Day 1, or unstable or uncontrolled condition (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
   2. Cardiac arrhythmia (Common Terminology Criteria for Adverse Events Grade 3 or higher) or clinically significant electrocardiogram (ECG) abnormalities
   3. ECG showing a baseline QT interval as corrected QTc >470 msec
5. Known:

   1. Active hepatitis A
   2. To be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen). Patients with resolved infection (i.e., patients who are positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.

      Exception: Patients with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
   3. To be seropositive for hepatitis C (except in the setting of a sustained virologic response, defined as aviremia at least 12 weeks after the completion of the antiviral therapy).
   4. Known to be seropositive for human immunodeficiency virus.
6. Patient has plasma cell leukemia (>2.0 × 109/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
7. Any concurrent medical or psychiatric condition or disease (e.g., active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results or that, in the opinion of the investigator, would constitute a hazard for participating in this study.
8. Ongoing ≥Grade 2 peripheral neuropathy.
9. Patient has had major surgery within two weeks before C1D1, or has not fully recovered from an earlier surgery, or has a surgery planned during the time the patient is expected to participate in the study or within two weeks after the last dose of study drug administration. Note: patients with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery.
10. Patient has known allergies, hypersensitivity, or intolerance to any of the study drugs, monoclonal antibodies, human proteins, or their excipients (refer to isatuximab Investigator's Brochure) or known sensitivity to mammalian-derived products.
11. Patient was vaccinated with live vaccines within four weeks prior to C1D1.
12. Pregnant or nursing women.
13. a. Females of childbearing potential (FCBP) unwilling to prevent pregnancy with the use of two reliable methods of contraception for ≥four weeks before the start of study treatment, during treatment (including dose interruptions), and up to five months following the last dose of isatuximab or three months following the last dose of the rest of the study treatment, whichever is longer. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap).

    b. FCBP who are unwilling or unable to be tested for pregnancy: a) twice before study treatment initiation (one 10-14 days prior to start of study drug and one within 24 hours prior to start of study drug. Urine tests must have a sensitivity of ≥25 mIU/mL), b) weekly during 1st month of treatment and then prior to each treatment cycle administration or c) every two weeks in case of irregular menstrual cycles, and d) up to five months following the last dose of isatuximab or three months following the last dose of the rest of the study treatment, whichever is longer.
14. Male participants who refuse to practice abstinence or use a condom during sexual contact with a pregnant female or an FCBP while participating in the study, during dose interruptions and at least five months following the last dose of isatuximab or three months following the last dose of the rest of the study treatment, whichever is longer, even if they have undergone a successful vasectomy.

Note 1: an FCBP is a female who: 1) has achieved menarche at some time point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Note 2: True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Renal Response Rate (RRR) | After six months of treatment with isatuximab plus VCd
  The primary endpoint is the renal response rate (RRR) after six months of treatment with isatuximab plus VCd. RRR is defined as the proportion of patients who achieve a partial renal (PRrenal) or better response after six months of treatment with isatuximab plus VCd, using the eGFR cut-off values of the IMWG response criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) | From study treatment initiation to progressive disease (PD), or initiation of further anti-myeloma treatment, or death, whichever comes first. Maximum time period 36 months
  The proportion of patients who achieve a partial response (PR) or better, assessed by the Investigator using the IMWG criteria, from study treatment initiation to progressive disease (PD), or initiation of further anti-myeloma treatment, or death, whichever comes first.
Progression-free survival (PFS) | From study treatment initiation to progressive disease (PD), or initiation of further anti-myeloma treatment, or death, whichever comes first. Maximum time period 36 months
  The time from study treatment initiation to the date of first documentation of PD, assessed by the Investigator using the IMWG response criteria, or initiation of further anti-myeloma treatment, or death from any cause, whichever comes first.
Time to Response (TTR) | From study treatment initiation to partial response (PR), or better. Maximum time period 36 months
  The time from study treatment initiation to the date of the first objective response of partial response (PR) or better, assessed with the IMWG response criteria.
Duration of Response (DoR) | From time response is achieved to progressive disease (PD), or death, whichever comes first. Maximum time period 36 months
  The time from the date of the first objective response to the date of the first documented PD, assessed by the Investigator using the IMWG response criteria, or death, whichever occurs first. DoR will be assessed only for patients who have achieved ≥ partial response (PR)
Overall Survival (OS) | From study treatment initiation to death. Maximum time period 36 months
  The time from study treatment initiation to the date of death from any cause. OS will be assessed during the response follow-up visits until the end of the study.
Minimal Residual Disease (MRD) negativity | Through study completion. Maximum time period 36 months
  The proportion of patients achieving MRD-negative status, assessed by the Investigator at suspected complete response as per IMWG criteria.
Safety Events i.e. Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs) and serious adverse events (SAEs) | Study treatment initiation until 30 days after last study treatment. Maximum time period 36 months
  The incidence of Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof, Principal Investigator — Department of Clinical Therapeutics, School of Medicine, National Kapodistrian University of Athens (NKUA)
Locations (6):
- Greece (6):
  - General Hospital of Athens "Evangelismos", Athens
  - Anticancer Oncology Hospital of Athens "Agios Savvas", Athens
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patra, Pátrai
  - Anticancer Hospital of Thessaloniki "Theageneio", Thessaloniki

IPD SHARING:
Plan to Share IPD: No